CLINICAL TRIAL: NCT04678024
Title: Multicentric Sensitivity Assessment of Antibody Diagnostic Tests Developed for Diagnosis of SARS-CoV2 Infection
Brief Title: Sensitivity Evaluation of Serological Tests for Covid-19
Acronym: COVIDIAGNOSTIX
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: COVIDIAGNOSTIX
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: test sierologici
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to test the diagnostic sensitivity of antibody tests for the diagnosis of SARS-CoV2 infection, available to clinical laboratories, within a national network of hospitals carrying out research activities. Test the diagnostic specificity of antibody tests for the diagnosis of SARS-CoV2 infection. Complete a systematic evaluation of the different approaches. Perform Health technology Assessment (HITA) of the methodologies under study, in order to verify their reliability to the immunoglobulin levels produced by each individual exposed patient.

ELIGIBILITY:
Inclusion Criteria:

All patients or individuals exposed to Sars-Cov2 Infection.

Exclusion Criteria:

There are no criteria for excluding patients or individuals, if not the refusal to participate to project

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients or individuals exposed to Sars-Cov2 Infection.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Up to 22 weeks
  Sensitivity and Specificity Evaluation in Diagnostic Sierological tests

SECONDARY OUTCOMES:
Specificity | Through study completion, an average of 1 year
  Sensitivity and Specificity Evaluation in Diagnostic Sierological tests

OTHER OUTCOMES:
HTA | Up to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Banfi, Principal Investigator — IRCCS Orthopedic Institute Galeazzi
Locations (1):
- Istituto Ortopedico Galeazzi, Milan, Italy